CLINICAL TRIAL: NCT06183424
Title: Effects of aTDCS Stimulation of the Dorsolateral Prefrontal Cortex on Cognitive Functions and the Parietal Memory Network, Default Mode Network in Patients Presenting Cognitive Symptoms After Covid-19 Infection: A Controlled Randomized Clinical Trial
Brief Title: TDCS Stimulation After Covid-19 Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Prof. Lutfu Hanoglu, MD, Prof. Dr. MD, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023IMU_ALKU_COVID
Record Dates: First submitted 2023-12-25; First posted 2023-12-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: Covid-19; tDCS; Cognitive function
MeSH Terms: conditions — COVID-19 | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Active Comparator): Active tDCS stimulation will be applied over the scalp for 20 minutes at an intensity of 2 mA. Stimulation will be given for 5 days. The application will be made to the patient who has had 30 Covid and has cognition complaints in a randomized manner.
  Interventions: Procedure: Transcranial Direct Stimulation
- Sham (Placebo Comparator): For the pseudo-stimulation to be applied to the sham group, the electrodes will be placed on the scalp in exactly the same way as the experimental group. For all stimulations, the reference electrode will be placed in the right orbital region and given once for 15 seconds, so that the participant will feel a slight tingling, but no real stimulation will be given.
  Interventions: Procedure: Transcranial Direct Stimulation

INTERVENTIONS:
Procedure: Transcranial Direct Stimulation — 2 mA, 20 min, 5 days

SUMMARY:
In this study, the effects of bilateral stimulation of the dorsolateral prefrontal cortex (DLPFC) with active tDCS (transcranial direct stimulation/transcranial direct stimulation) on neurocognitive (memory and executive) functions in patients with Covid-19 infection and subjective cognitive complaints, as well as resting-state fMRI In the case of dfMRI, it is aimed to examine the default mode network (DMN) and parietal memory network (PMN) inter- and intra-network connectivity alterations and the hippocampal region connectivity alterations and contribute to the relevant literature.

DETAILED DESCRIPTION:
The DMN is active when not engaged in a goal-oriented activity and at rest. Resting DNM is especially active when the mind is busy with introspective situations (Barkhof et al., 2014; Mak et al., 2017). Although the posterior parts of the DMN consisting of the posterior cingulate/precuneus and bilateral parietal cortex regions are associated with memory functions, memory functions are not unique to DMN and the parietal regions are not functionally homogeneous (Sestieri et al., 2011). At this point, a new network called the parietal memory network (PMN) was defined in a study by Gilmore (Gilmore et al., 2015). This network is a system that diverges from the posterior parts of the DMN and consists of the middle cingulate cortex, precuneus and inferior parietal lobule/angular gyrus structures and has overlapping regions with the DMN. This network appears to differ from the DMN in different types of recall memory functions. Accordingly, when recalling autobiographical information, DMN; PMN seems to be active in encoding and recall tasks related to recognition memory (McDermott et al., 2009; Chen et al., 2017; Nelson et al., 2013; Hu et al., 2016; Manenti et al., 2010; Kragel et al., 2016) . A double dissociation appears to occur between these two network systems in memory processes, and furthermore, the spacial proximity of PMN to the DMN suggests that some of the cognitive dysfunctions attributed to the DMN of these two systems are due to PMN. The fact that PMN is associated with memory encoding and recall functions even in different types of tasks (de-activity in perceiving new stimulus but being active in perceiving familiar stimulus) differentiates it from other network systems. Stimulation of the parietal region with repetitive transcranial magnetic stimulation (rTMS) resulted in improved visual recognition memory performance (Velioğlu et al., 2021).

The dorsolateral prefrontal cortex (DLPFC) is the central region associated with executive functions, and damage to this region is associated with difficulty in regulating behavioral responses, memory-retrieval, and inability to demonstrate appropriate motor behavior. Damages in this region are associated with cognitive loss in related areas (Liu et al., 2021; Brak et al., 2022). tDCS, on the other hand, stands out as a promising method for patients with Covid-19 infection and subjective cognitive complaints, and appears to act by modulating functional connectivity (Baptista, 2020; Linnhoff, 2023; Yulug B). Increased connectivity between the hippocampus and other DMN nodes such as the dorsal attention network, control, attention-attractiveness network, and sensori-motor networks was detected in fMRI with atDCS stimulation (Manenti et al., 2020; Meinzer et al., 2015). In this context, improvement in neurocognitive tests and changes in functional imaging can be detected with stimulation of the relevant regions of the cortex with tDCS in patients who have had Covid-19 infection and have subjective cognitive complaints. In patients with Covid-19 infection, stimulation of the relevant regions with tDCS resulted in improvement in cognitive functions such as working memory and cognitive control. (Baptista, 2020; Linnhoff, 2023; Yulug B,2023). At this point, DLPFC stimulation may also result in improved cognitive functions regarding encoding and recall.

From this point of view, in this study -based on the studies referenced in the text-, bilateral stimulation of the DLPFC region with anodal tDCS (atDCS) increased performance in neurocognitive abilities, especially memory and executive functions, in patients who had Covid-19 infection and had subjective cognitive complaints. The methodical mesh is shaped in the context of this template, hypothesizing that it will result in In addition, in the fMRI studies mentioned above, it is aimed to point out that tDCS stimulation increases the coherence between DMN networks and to examine the effect of tDCS stimulation on DMN network connectivity and connectivity with the hippocampal region with reference to the role of PMN in patients with Covid-19 infection and subjective cognitive complaints. From this point of view, the aim of this study is dorsolateral prefrontal cortex (DLPFC) active tDCS (transcranial direct stimulation/transcribed) in patients with covid-19 infection and subjective cognitive complaints.

ELIGIBILITY:
Inclusion Criteria:

* Have received a positive value from the COVID-19 RT-PCR test in the last 60 days and turned negative
* Being between the ages of 18-50
* 21 days have passed since the disease onset date

Exclusion Criteria:

* Having any neurological or psychiatric disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment | Before Treatment / 1 month after treathment
  Cognition Test
Cognition Test Material | Before Treatment / 1 month after treathment
  clock drawing test, digit range test, verbal fluency test, stroop test, trail making test
NPI | Before Treatment / 1 month after treathment
  Cognition Test (Neuropsychiatric Inventory)
Öktem Verbal Memory Processes Test | Before Treatment / 1 month after treathment
  Cognition Test
Rey Complex Figure Test | Before Treatment / 1 month after treathment
  Cognition Test

CONTACTS AND LOCATIONS:
Overall Officials: Burak Yuluğ, Prof. DR. MD, Study Director — Alanya Alaaddin Keykubat Üniversitesi
Locations (1):
- Alanya Alaaddin Keykubat Üniversitesi, Antalya, Turkey (Türkiye)